CLINICAL TRIAL: NCT00478725
Title: An Open-Label, Two-Part Study to Characterize the Pharmacokinetics of a Single Intravenous Dose of Pazopanib (GW786034) and the Absorption, Distribution, Metabolism and Elimination of a Single Oral [14C] Labeled Dose of Pazopanib in Subjects With Solid Tumor Malignancies
Brief Title: Part A: Radiolabel Study With GW786034 Part B: Single Dose of GW786034
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEG10004
Record Dates: First submitted 2007-05-24; First posted 2007-05-25 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Carcinoma, Renal Cell
Keywords: Metastatic Cancer; Advanced Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Absorption, Distribution, Metabolism and Elimination of a Single Oral [14C] Labeled Dose of GW786034
  Interventions: Drug: GW786034, oral; Drug: GW786034, radiolabeled oral
- Part B (Experimental): characterize the pharmacokinetics of a single IV dose of GW786034
  Interventions: Drug: GW786034, oral; Drug: GW786034, IV

INTERVENTIONS:
Drug: GW786034, oral — oral, 800 mg
  Other Names: GW786034; pazopanib
Drug: GW786034, IV — IV, 5 mg
  Other Names: GW786034; pazopanib
  Arms: Part B
Drug: GW786034, radiolabeled oral — oral, 400 mg radiolabeled
  Other Names: GW786034; pazopanib
  Arms: Part A

SUMMARY:
To study the absorption, distribution, metabolism and excretion of GW786034, and the absorption of a single IV dose of GW786034

ELIGIBILITY:
Inclusion criteria:

* Subject must provide written informed consent prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow-up. Procedures conducted as part of the subject's routine clinical management (e.g., blood count, imaging study) and obtained prior to signing of informed consent may be utilized for screening or baseline purposes provided these procedures are conducted as specified in the protocol.
* Has histologically or cytologically confirmed advanced solid tumor malignancy.
* For Part A: Males, age: 30 years or greater.
* For Part B: Males or Females, age: 18 years or greater.
* For Part A or B, males that meet the following criteria.
* A male subject with a female partner of childbearing potential is eligible to enter and participate in this study if he:

  * Agrees to use double-barrier contraception (condom with spermicidal jelly, foam, suppository or film, or a condom and his partner uses a diaphragm with spermicide), OR
  * Agrees to complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the clinical trial, and for at least 21 days after the last dose of investigational product.
* For Part B, females that meet the following criteria:
* A female subject is eligible to enter and participate in this study if she is of:

  * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had:

    * A hysterectomy
    * A bilateral oophorectomy (ovariectomy)
    * A bilateral tubal ligation
    * Is post-menopausal (total cessation of menses for >/ 1 year), OR
  * Childbearing potential and has a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception. GSK acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follows:

    * An intrauterine device (IUD) with a documented failure rate of less than 1% per year.
    * Vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
    * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the clinical trial, and for at least 21 days after the last dose of investigational product.
    * Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide).
* Note: Oral contraceptives are not considered reliable due to potential drug-drug interaction.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Body weight >/ 50 kg.
* Adequate organ systems function as defined in Table 1.
* Ability to swallow and retain oral medication.

Exclusion criteria:

* History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to beginning study treatment. Screening with CNS imaging studies (CT scan or MRI) is required only if clinically indicated or if the subject has a history of CNS metastases.
* Clinically significant gastrointestinal (GI) abnormalities including, but not limited to: malabsorption syndrome, history of resection of the stomach or small bowel, active peptic ulcer disease, inflammatory bowel disease, ulcerative colitis or other conditions that increase the risk for perforation, history of abdominal fistula, GI perforation or intra-abdominal abscess within 4 weeks prior to beginning study treatment.
* Presence of uncontrolled infection.
* Corrected QT interval (QTc) > 480 msec.
* History of any one or more of the following cardiovascular conditions within the past 6 months: congestive heart failure, cardiac angioplasty or stenting, myocardial infarction, unstable angina OR symptomatic peripheral vascular disease.
* Has poorly controlled hypertension (systolic blood pressure [SBP] >/ 140 mmHg, or diastolic blood pressure [DBP] >/ 90 mmHg).
* Note: Initiation or adjustment of anti-hypertensive medication(s) is permitted prior to study entry. The blood pressure (BP) must be re-assessed on 2 occasions that are separated by a minimum of 24 hours. The mean SBP/DBP values from both BP assessments must be < 140/90 mmHg in order for a subject to be eligible for the study.
* History of cerebrovascular accident or pulmonary embolism within the past 6 months.
* History of untreated deep venous thrombosis (DVT) within the past 6 months.
* Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible.
* Prior major surgery or trauma within the past 28 days or presence of any wound, fracture or ulcer which is not fully healed.
* Evidence of active bleeding, bleeding diathesis or hemoptysis within 6 weeks prior to study treatment.
* Use of prohibited medications within the timeframes specified in Section 9.2, Prohibited Medications of the protocol.
* Use of an investigational agent, including an investigational anti-cancer agent within 28 days or 5 half-lives, whichever is longer, preceding the first dose of pazopanib.
* Treatment with any cancer therapy (including chemotherapy, radiation therapy, immunotherapy, biologic therapy, hormonal therapy, surgery or tumor embolization) within 14 days prior to the first dose of pazopanib.
* Note: Current treatment with leuprolide is permitted.
* Any ongoing potentially reversible toxicity from prior anti-cancer therapy that is > Grade 1 or any toxicity from prior anti-cancer therapy that is progressing in severity.
* Any serious and/or unstable pre-existing medical, psychiatric, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study, including any condition that could interfere with the accurate assessment and recovery of [14C].
* History or presence of hepatic or renal disease or any other condition known to interfere with the absorption, distribution, metabolism or excretion of drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-07-18 (Actual); Primary Completion 2008-07-01 (Actual); Study Completion 2008-07-01 (Actual)

PRIMARY OUTCOMES:
Part A: excretion of radioactivity | over 168 hrs
Part B: Plasma pazopanib, clearance (CL) and AUC(0-t), AUC(0-8),Cmax and half-life (t1/2) pazopanib and pazopanib metabolites (GSK 1268992, GSK1268997, GSK1071306 and GW700201) | over 48 hrs

SECONDARY OUTCOMES:
Part A: Blood and plasma total radioactivity AUC(0-t), AUC(0-8),Cmax and t1/2 | over 168 hrs.
Part B: Safety parameters | over 48 hrs.
Blood and plasma total radioactivity AUC(0-t), AUC(0-∞), Cmax and t1/2 following oral administration of 400 mg of [14C]-pazopanib containing approximately 70 µCi of radioactivity. | on Day 15 of Cycle 1.
Samples (for use in a separate study) to characterize and quantify metabolites of pazopanib in plasma, urine and feces. | on Day 15 of Cycle 1.
Blood:plasma ratio of total drug-related material (radioactivity). | on Day 15 of Cycle 1.
Plasma pazopanib AUC(0-t), AUC(0-∞), Cmax, tmax following oral administration of 400 mg of [14C]-pazopanib containing 70 µCi of radioactivity. | on Day 15 of Cycle 1.
Safety parameters: adverse events (AEs), vital signs, electrocardiograms (ECGs) and clinical laboratory assessments. | on Day 15 of Cycle 1.
Plasma pazopanib AUC(0-24), Cmax, tmax following oral administration of 800 mg pazopanib | on Day 15 of Cycle 1.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Nashville, Tennessee

REFERENCES:
- [Background] Deng Y, Sychterz C, Suttle AB, Dar MM, Bershas D, Negash K, Qian Y, Chen EP, Gorycki PD, Ho MY. Bioavailability, metabolism and disposition of oral pazopanib in patients with advanced cancer. Xenobiotica. 2013 May;43(5):443-53. doi: 10.3109/00498254.2012.734642. Epub 2012 Nov 16. PMID 23548165
- See also: Results for study VEG10004 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/VEG10004?search=study&search_terms=VEG10004#rs